CLINICAL TRIAL: NCT01247025
Title: Examining Prolonged Grief Disorder and Its Relationship to Self-Directed Violence Among Veterans
Brief Title: Prolonged Grief and Suicide Among Veterans
Status: Withdrawn | Type: Observational
Why Stopped: Study should not have been listed on ClinicalTrials.gov
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Peter M. Gutierrez, Ph.D./ Clinical research Psychologist, VA VISN 19 MIRECC
Other Study IDs: jrings1
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Prolonged Grief Disorder; Suicidality
MeSH Terms: conditions — Prolonged Grief Disorder; Suicidal Ideation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Veterans: Veterans receiving mental health services at the Eastern Colorado Healthcare System (ECHCS)/Denver Veterans Affairs Medical Center (VAMC)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study will not contain a specific intervention

SUMMARY:
The primary research question in this study will ask, among those receiving outpatient mental health services (MHS) at the Eastern Colorado Healthcare System (ECHCS)/Denver Veterans Affairs Medical Center (VAMC), how many suffer from Prolonged Grief Disorder (PGD)? Here, it is hypothesized that PGD will occur within the sample. A secondary aim of this study will be to investigate how often PGD co-occurs with posttraumatic stress disorder (PTSD) and/or depression. Also, while PGD has been shown to have an effect on self-directed violence (SDV) among civilians (Prigerson, Bridge et al., 1999), no studies yet have examined the relationship between PGD and SDV among Veterans. Therefore, it also is hypothesized that as PGD severity increases among the Veteran sample, risk for SDV will increase as well. Additional research aims also will be addressed in this study. For one, it will be assessed which grief symptoms are most often reported among the Veteran sample. Also, no study has yet to examine if there are neuropsychological differences between PGD and PTSD. Therefore, another research question here is whether PGD indeed is neuropsychologically different from PTSD. Here, the exploratory hypothesis is that PGD sufferers will respond to a measure of multiple components of cognition (e.g., planning, sequencing, concentration, multitasking, and memory efficiency) in a manner that is significantly different from PTSD sufferers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Not currently active duty in any branch of the military
* English-speaking
* Ability to adequately respond to specific questions regarding the informed consent procedure.
* Active case in Mental Health Services (MHS) at the Eastern Colorado Healthcare System (ECHCS)/Denver Veterans Affairs Medical Center (VAMC)

Exclusion Criteria:

* Currently active duty in any branch of the military
* Non-English-speaking
* Inability to adequately respond to questions regarding the informed consent procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants in this observational study will be all individuals willing and eligible among those seeking outpatient mental health services at the Eastern Colorado Healthcare System (ECHCS)/Denver Veterans Affairs Medical Center (VAMC). It is expected that 180 participants will be enrolled in an effort to obtain up to 150 completed protocols. Women and minorities will be recruited as a routine part of the study. However, given the participant population within the Eastern Colorado Healthcare System (ECHCS)/Denver Veterans Affairs Medical Center (VAMC), it is expected the majority of participants will be Caucasian men.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Prolonged Grief Disorder- 13 | At least six months post-bereavement

SECONDARY OUTCOMES:
Adult Suicidal Ideation Questionnaire | Within past month

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Gutierrez, PhD, Principal Investigator — VA Eastern Colorado Health Care System
Locations (2):
- United States (2):
  - Eastern Colorado Health Care System (ECHCS) / Denver VA Medical Center, Denver, Colorado
  - VA Eastern Colorado Health Care System, Denver, Colorado